CLINICAL TRIAL: NCT03704532
Title: Nonoperative Treatment of Acute Achilles Tendor Rupture in Central Finland: Prospective Cohort Study
Brief Title: Nonoperative Treatment of Acute Achilles Tendor Rupture
Acronym: NoArc
Status: Active, not recruiting | Type: Observational
Sponsor: Central Finland Hospital District (Other)
Collaborators: University of Jyvaskyla (Other)
Responsible Party: Sponsor
Other Study IDs: 2U/2018
Record Dates: First submitted 2018-10-10; First posted 2018-10-12 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Achilles Tendon Rupture
Keywords: achilles tendon rupture; nonoperative treatment; functional rehabilitation; operative treatment; biomechanical measurements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Operative treatment: Patients having undergone an operative treatment of achilles tendon rupture
  Interventions: Procedure: Operative treatment
- Nonoperative treatment: Patients having undergone a nonoperative treatment with functional rehabilitation of achilles tendon rupture
  Interventions: Procedure: Nonoperative treatment

INTERVENTIONS:
Procedure: Operative treatment — Open surgical repair of tendon rupture
  Groups: Operative treatment
Procedure: Nonoperative treatment — Nonoperative treatment with lower leg orthosis and functional rehabilitation
  Groups: Nonoperative treatment

SUMMARY:
A prospective, non-randomised, observational study to investigate the clinical and biomechanical outcomes and prevalence of reruptures after operative or nonoperative treatment of acute achilles tendon rupture.

ELIGIBILITY:
Inclusion Criteria:

* acute achilles tendon rupture with clear onset of symptoms
* closed rupture
* resides in the catchment area of our hospital district

Exclusion Criteria:

* avulsion fractures in the calcaneus
* unwillingness to participate
* inability to communicate using Finnish language

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients having sustained an acute achilles tendon rupture and referred for either operative or nonoperative treatment with functional rehabilitation at our institution.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rerupture rate | 1 year
  Rate rerupture of a healed tendon after the end of the intervention

SECONDARY OUTCOMES:
Physical Activity Level | 1 year
  Patient activity 1 year after the rupture using the Tegner activity level scale which varies from 0 to 10. This scale that aims to provide a standardized method of grading work and sporting activities.
University of California, Los Angeles (UCLA) score | 1 year
  Patient activity 1 year after the rupture
Achilles tendon rupture score (ATRS) | 1 year
  Achilles tendon rupture score 1 year after the rupture
Functional Score | 1 year
  Leppilahti score measuring subjective and objective functional outcome 1 year after the rupture on a scale 0-100.
Foot inversion | 1 year
  Foot inversion angle in rest
Foot flexion-extension | 1 year
  Foot flexion-extension angle in rest
Heel-raise test | 1 year
  One leg heel-raise test while standing

OTHER OUTCOMES:
Muscle strength | 1 year
  Isometric plantar flexion strength
Gastrocnemius muscle cross-sectional area | 1 year
  Lateral and medial gastrocnemius and soleus muscle area using ultrasound
Tendon length | 1 year
  Achilles tendon length using ultrasound
Research ANd Development (RAND-36) quality of life | 1 year
  Measurement of quality of life using RAND-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Juha Paloneva, MD, PhD, Study Chair — Central Finland Health Care District
Locations (1):
- Central Finland Hospital, Jyväskylä, Central Finland, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sukanen M, Khair RM, Reito A, Ponkilainen V, Paloneva J, Cronin N, Hautala AJ, Finni T. Early Predictors of Recovery From Nonoperatively Treated Achilles Tendon Rupture: 1 Year Follow-Up Study. Scand J Med Sci Sports. 2024 Jul;34(7):e14700. doi: 10.1111/sms.14700. PMID 39010659